CLINICAL TRIAL: NCT07271836
Title: Effect of Structured Counseling on Continuation Rates of Long Acting Reversible Contraception Among Clients Requesting Early Removal: A Multicenter Randomized Controlled Trial (PLACE Trial)
Brief Title: PLACE Trial: Preserving Long-Acting Contraception Through Education
Acronym: PLACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Muhammad Ibrahim Khan, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSAIRB
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Contraception
Keywords: long acting reversible contraception; LARC; subdermal implant; jadelle; intrauterine contraceptive device; copper-t; counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured counseling (Experimental): Women in this arm will receive structured, culturally sensitive counseling by trained healthcare providers. The counseling aims to address common myths and misconceptions about long-acting reversible contraception (LARC), such as concerns about side effects (e.g., amenorrhea, pregnancy worries) and general fears related to the method. The goal is to encourage continued use of LARC unless women meet the WHO criteria for removal (e.g., medical complications or personal preference). Participants will be followed up for 6 months to assess if they continue using their LARC method.
  Interventions: Behavioral: Structured counseling
- No counseling (No Intervention): Women in this arm will receive standard care, which is the typical practice at the clinics. If they request to remove their contraceptive device (either a copper-T IUD or Jadelle implant), it will be removed upon request without any counseling or encouragement to continue the method. There will be no structured intervention. Participants will not be asked to follow-up after the initial visit.

INTERVENTIONS:
Behavioral: Structured counseling — The intervention is a behavioral intervention where healthcare providers deliver structured, culturally sensitive counseling to women who present for early removal of their long-acting reversible contraception (LARC), such as the copper-T intrauterine device (IUD) or Jadelle subdermal implant. The counseling is designed to address common misconceptions and myths about contraception, such as fears related to side effects (e.g., amenorrhea, concerns about pregnancy) or the belief that symptoms are unrelated to the contraception method. The aim is to encourage the continuation of the contraceptive method unless the woman meets the WHO criteria for removal (e.g., medical reasons or personal preference). This intervention will involve a one-time counseling session with follow-up at 6 months to assess whether the participant continued or discontinued the method.
  Arms: Structured counseling

SUMMARY:
Study Overview Summary

This randomized controlled trial will evaluate the effectiveness of structured counseling in improving the continuation rates of long-acting reversible contraception (LARC) among women in Islamabad, Pakistan, who present to family planning clinics for early removal of their contraception devices (copper-T IUD or Jadelle implant). The study, starting December 15, 2025, will recruit women from three federal government-approved clinics.

The trial will randomly assign participants to either an intervention group, where they will receive culturally sensitive counseling to encourage continued use of LARC, or a control group, where contraception will be removed upon client request without counseling. The goal is to determine if structured counseling can increase the likelihood of women continuing their LARC method.

DETAILED DESCRIPTION:
Study Overview

This randomized controlled trial aims to assess the effectiveness of structured counseling on the continuation rates of long-acting reversible contraception (LARC) among women who present to family planning clinics in Islamabad, Pakistan, for early (within two years of use) removal of their contraception devices. The study will specifically target women who seek to remove either the copper-T intrauterine contraceptive device (IUD) or the Jadelle subdermal implant.

Starting December 15th, 2025, the research team will recruit eligible participants from three major federal government-approved family planning clinics in Islamabad. The clinics will serve as the intervention and control settings, with half of the healthcare providers trained in a standardized, culturally sensitive counseling approach, while the other half will provide standard care by simply removing the contraceptive device upon request.

The trial will aim to determine whether structured counseling can effectively increase the likelihood of women continuing with their LARC method as compared to the control group, where no counseling intervention is provided.

Study Design

This is a multicenter, randomized controlled trial with a parallel-group design conducted across three family planning clinics in Islamabad, Pakistan. The study will randomly assign participants to one of two groups:

Intervention and Control Groups (Please refer to the 'arms and interventions' pane for details).

The intervention group will also be followed up for 6 months post-visit either in clinic or via teleconsultation to assess the continuation of the contraception method.

Recruitment and Randomization

Recruitment: Starting December 15, 2025 for the first two months, women will be recruited from the family planning clinics when they present for the removal of either a copper-T IUD or a Jadelle implant that has been in place for 2 years or less. Participants who do not meet the inclusion criteria (e.g., not presenting within the first two months of start of the study) will be excluded. Informed written consent will be taken from each client and clients asked to fill a questionnaire.

Randomization: Women will be randomly assigned to either the intervention group (structured counseling) or the control group (standard care). Randomization will be performed using a computer-generated randomization scheme. Each participant will be assigned a unique clinic visit slip that indicates the assigned group (intervention or control) and specifies the clinic room number.

Provider Training

Intervention Group: Healthcare providers at each of the three clinics will receive training on standardized counseling techniques, focusing on culturally sensitive approaches. The training will cover topics such as addressing questions, common myths and misconceptions about LARC, such as fears related to amenorrhea, concerns about pregnancy, and misattributions of symptoms unrelated to contraception. The aim of the counseling will be to encourage clients to continue their contraception method, provided they do not meet the WHO criteria for removal (e.g., medical complications, side effects, or personal preference).

After the training, feedback and detailed assessments of the providers will be conducted to ensure provider bias is minimized and that the counseling is delivered as per the protocol.

Control Group: The remaining providers at the clinics will not receive any training on counseling. These providers will be instructed to remove the contraceptive device upon client request without providing any counseling or intervention to encourage continuation. However, clients will be asked to complete a questionnaire to help analyze the reasons for contraceptive removal, which will be used to assess the potential impact of counseling on the continuation of the LARC method.

Sample Size Calculation

The sample size was calculated based on the contraceptive prevalence rate for Pakistan, which is approximately 34%. The expected effect size is a 30% difference in continuation rates between the intervention and control groups. The 95% confidence interval and a 5% margin of error were used to calculate the required sample size. A statistical power of 90% was used. Furthermore, an anticipated 50% loss to follow-up was factored into the sample size calculation.

For each contraceptive method (IUD or implant) and each clinic, the sample size for both arms (intervention and control) is estimated to be 49 participants per method, per clinic. Therefore, the total sample size for all three clinics, across both arms and methods, is calculated to be 588 participants. To account for potential record losses, the sample size has been increased by 50%, bringing the total required sample size to 900 participants (300 participants per center).

Statistical Analysis

Statistical analysis will compare the continuation rates of LARC between the intervention group (structured counseling) and the control group (standard care) using an intention-to-treat approach. Descriptive statistics will be used to summarize demographic data, and Chi-square tests will be used to compare proportions of women continuing contraception in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting at the clinics exclusively for removal of a copper-T IUD or Jadelle subdermal implant within 2 years of use and within the first 2 months of the study.

Exclusion Criteria:

* Women not wishing to participate or unable to provide informed consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females only.
Enrollment: 900 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Continuation Rate of Long-Acting Reversible Contraception (LARC) at 6 Months | The total study duration will be eight months: the first two months will be allocated to enrolling participants and completing their baseline visits, followed by a six-month follow-up period for all enrolled clients.
  The primary outcome of the study is the rate of LARC continuation in women who received either structured counseling (intervention arm) or standard care (control arm) for the continuation of their intrauterine contraceptive device (IUD) or subdermal implant (Jadelle). The continuation rate will be assessed at a 6-month follow-up after the initial clinic visit.
  Intervention Group: Participants who receive structured, culturally sensitive counseling will be encouraged to continue using their LARC method unless they meet the WHO criteria for removal (e.g., medical complications, side effects, or personal preference).
  Control Group: Participants in the control group, who receive standard care (removal of the device upon request without any counseling), will be asked to return for a 6-month follow-up to determine if they have continued or discontinued their contraception method.
  Unit of measurement: Percentage of women that continued the chosen method following the visit.

SECONDARY OUTCOMES:
Client Satisfaction and Factors Influencing Contraceptive Continuation | Eight months
  The secondary outcomes of this study aim to assess client satisfaction with the LARC method.
  Client Satisfaction: At the 6-month follow-up, participants will be asked to complete a brief survey or interview assessing their overall satisfaction with the contraception method they are using (IUD or subdermal implant). This will include questions about the comfort, effectiveness, and side effects of the method, as well as their level of confidence in the method.
  Unit of measurement: Likert scale score (1-5, where 1 = very unsatisfied and 5 = very satisfied)
Factors Influencing Contraceptive Continuation | Eight months
  Another secondary outcome is to identify the factors influencing the decision to continue or discontinue the contraceptive method, focusing on those who received structured counseling (intervention group) and those who received standard care (control group).
  The study will gather detailed information on the reasons for discontinuation or continuation of the LARC method. This includes identifying specific concerns related to side effects-such as amenorrhea, irregular or heavy bleeding, cramping, discomfort, weight changes, and perceived hormonal effects-as well as fears rooted in myths and misconceptions (e.g., infertility, device migration, long-term health risks).
  Unit of measurement: Categorical variables e.g. amenorrhea with frequency counts.

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Rhs 'A' Center Federal Government Poly Clinic (Fgpc), Islamabad, Islamabad
  - RHS 'A' CENTER Mother and Child Health Centre Aabpara, Islamabad, Islamabad
  - RHS-A centre, Pakistan Institute of Medical Sciences, Islamabad, Islamabad

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including demographics, clinical outcomes, and adverse events, will be available beginning 6 months after publication of the primary results. Data will be shared through a controlled-access repository to qualified researchers upon request and after signing a data use agreement
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From August 2026 onwards

REFERENCES:
- [Background] Gibbs SE, Rocca CH, Bednarek P, Thompson KMJ, Darney PD, Harper CC. Long-Acting Reversible Contraception Counseling and Use for Older Adolescents and Nulliparous Women. J Adolesc Health. 2016 Dec;59(6):703-709. doi: 10.1016/j.jadohealth.2016.07.018. Epub 2016 Sep 21. PMID 27665153